CLINICAL TRIAL: NCT04619511
Title: Risk Factors for Post-ESWL and Post-ERCP Pancreatitis in Patients With Chronic Pancreatitis
Brief Title: Risk Factors for Post-ESWL and Post-ERCP Pancreatitis
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Principal Investigator, Changhai Hospital
Other Study IDs: ESWL&ERCP
Record Dates: First submitted 2020-11-03; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pancreatitis; Risk Factors; ERCP; ESWL
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aimed to identify risk factors for post-ERCP pancreatitis(PEP) after ESWL, and the relationship between the occurrence of post-ESWL pancreatitis and PEP.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic pancreatitis and treated with both ESWL and subsequent ERCP

Exclusion Criteria:

* Patients with isolated pancreatic tail stone
* Patients with suspected or established malignancy
* Patients with pancreatic ascites
* Patients attending other interventional clinical trials
* Patients with non-correctable coagulation disorder
* Patients with pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive CP patients treated with both ESWL and subsequent ERCP during the same hospitalization between October 2016 and July 2019 were included.
Sampling Method: Non-Probability Sample
Enrollment: 714 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
post endoscopic retrograde cholangiopancreatography(ERCP) pancreatitis | up to 1 months
  The main outcome analyzed was the development of post-procedural pancreatitis, which was defined as clinical pancreatitis, meeting two of three the following criteria in accordance with the Revised Atlanta International consensus including pain consistent with AP; amylase or lipase more than 3 times the upper normal limit; characteristic findings on imaging.
post pancreatic extracorporeal shock wave lithotripsy (ESWL) pancreatitis | up to 1 months
  The main outcome analyzed was the development of post-procedural pancreatitis, which was defined as clinical pancreatitis, meeting two of three the following criteria in accordance with the Revised Atlanta International consensus including pain consistent with AP; amylase or lipase more than 3 times the upper normal limit; characteristic findings on imaging.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ru N, Qian YY, Zhu JH, Chen H, Zou WB, Hu LH, Pan J, Guo JY, Li ZS, Liao Z. Post-ESWL and post-ERCP pancreatitis in patients with chronic pancreatitis: Do they share the same risks? J Hepatobiliary Pancreat Sci. 2021 Sep;28(9):778-787. doi: 10.1002/jhbp.1013. Epub 2021 Jul 22. PMID 34242478